CLINICAL TRIAL: NCT04857554
Title: Effects of Sugar-free Products With Added Sweeteners: Apricot Jam, Cranberry Cereal Bar, and Cocoa Drink on Glycemic Responses: Randomized Clinical Trial in Healthy Humans
Brief Title: Effects of Sugar-free Products With Added Sweeteners on Glycemic Responses
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Agricultural University of Athens (Other)
Responsible Party: Principal Investigator, Aimilia Papakonstantinou, Assistant Professor, Agricultural University of Athens
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Other
Other Study IDs: HRBD 23 08/07/2020
Record Dates: First submitted 2021-04-21; First posted 2021-04-23 (Actual); Last update posted 2021-04-23 (Actual); Status verified 2021-04

CONDITIONS: Potential Abnormality of Glucose Tolerance; Appetitive Behavior
Keywords: blood glucose; glycemic index; cereal bar; jam; cocoa
MeSH Terms: conditions — Appetitive Behavior | interventions — Glucose

STUDY DESIGN:
Intervention Model Description: Crossover Assignment
Who Masked: Investigator
Masking Description: Single (Investigator)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- Glucose as reference food (Experimental): Twelve healthy, normal weight subjects (male: 6, female: 6) after 10-14 hr fast, consumed 25g available carbohydrate from D-glucose, three times, in different weeks as reference food along with 250ml water; and 25g available carbohydrates from white bread, white bread and apricot jam, cereal bar with cranberries, and cocoa drink, tested once, in different weeks along with 250ml water or 500ml fat-free milk for the cocoa drink. Fingertip capillary blood glucose samples were taken at baseline, 15, 30, 45, 60, 90 and 120min. The first glucose sample was taken exactly 15min after the first bite of food or drink.
  Interventions: Other: Glucose as reference food; Other: White bread as reference food; Other: White bread with apricot jam; Other: Cereal bar with cranberries; Other: Cocoa drink
- White bread as reference food (Experimental): Twelve healthy, normal weight subjects (male: 6, female: 6) after 10-14 hr fast, consumed 25g available carbohydrate from D-glucose, three times, in different weeks as reference food along with 250ml water; and 25g available carbohydrates from white bread, white bread and apricot jam, cereal bar with cranberries, and cocoa drink, tested once, in different weeks along with 250ml water or 500ml fat-free milk for the cocoa drink. Fingertip capillary blood glucose samples were taken at baseline, 15, 30, 45, 60, 90 and 120min. The first glucose sample was taken exactly 15min after the first bite of food or drink.
  Interventions: Other: Glucose as reference food; Other: White bread as reference food; Other: White bread with apricot jam; Other: Cereal bar with cranberries; Other: Cocoa drink
- White bread with apricot jam (Experimental): Twelve healthy, normal weight subjects (male: 6, female: 6) after 10-14 hr fast, consumed 25g available carbohydrate from D-glucose, three times, in different weeks as reference food along with 250ml water; and 25g available carbohydrates from white bread, white bread and apricot jam, cereal bar with cranberries, and cocoa drink, tested once, in different weeks along with 250ml water or 500ml fat-free milk for the cocoa drink. Fingertip capillary blood glucose samples were taken at baseline, 15, 30, 45, 60, 90 and 120min. The first glucose sample was taken exactly 15min after the first bite of food or drink.
  Interventions: Other: Glucose as reference food; Other: White bread as reference food; Other: White bread with apricot jam; Other: Cereal bar with cranberries; Other: Cocoa drink
- Cereal bar with cranberries (Experimental): Twelve healthy, normal weight subjects (male: 6, female: 6) after 10-14 hr fast, consumed 25g available carbohydrate from D-glucose, three times, in different weeks as reference food along with 250ml water; and 25g available carbohydrates from white bread, white bread and apricot jam, cereal bar with cranberries, and cocoa drink, tested once, in different weeks along with 250ml water or 500ml fat-free milk for the cocoa drink. Fingertip capillary blood glucose samples were taken at baseline, 15, 30, 45, 60, 90 and 120min. The first glucose sample was taken exactly 15min after the first bite of food or drink.
  Interventions: Other: Glucose as reference food; Other: White bread as reference food; Other: White bread with apricot jam; Other: Cereal bar with cranberries; Other: Cocoa drink
- Cocoa drink (Experimental): Twelve healthy, normal weight subjects (male: 6, female: 6) after 10-14 hr fast, consumed 25g available carbohydrate from D-glucose, three times, in different weeks as reference food along with 250ml water; and 25g available carbohydrates from white bread, white bread and apricot jam, cereal bar with cranberries, and cocoa drink, tested once, in different weeks along with 250ml water or 500ml fat-free milk for the cocoa drink. Fingertip capillary blood glucose samples were taken at baseline, 15, 30, 45, 60, 90 and 120min. The first glucose sample was taken exactly 15min after the first bite of food or drink.
  Interventions: Other: Glucose as reference food; Other: White bread as reference food; Other: White bread with apricot jam; Other: Cereal bar with cranberries; Other: Cocoa drink

INTERVENTIONS:
Other: Glucose as reference food — Twelve healthy, normal weight subjects (male: 6,female: 6) after 10-14 hr fast, consumed 25g glucose diluted in 250ml water, tested twice, in different weeks, within 5-10min. Fingertip capillary blood glucose samples were taken at baseline, 15, 30, 45,60, 90 and 120min.
Other: White bread as reference food — Twelve healthy, normal weight subjects (male: 6,female: 6) after 10-14 hr fast, consumed 25g available carbohydrates from white bread along with 250ml water, tested once, in different weeks, within 10-15min. Fingertip capillary blood glucose samples were taken at baseline, 15, 30, 45,60, 90 and 120min.
Other: White bread with apricot jam — Twelve healthy, normal weight subjects (male: 6,female: 6) after 10-14 hr fast, consumed 25g available carbohydrates from white bread together with apricot jam along with 250ml water, tested once, in different weeks, within 10-15min. Fingertip capillary blood glucose samples were taken at baseline, 15, 30, 45,60, 90 and 120min.
Other: Cereal bar with cranberries — Twelve healthy, normal weight subjects (male: 6,female: 6) after 10-14 hr fast, consumed 25g available carbohydrates from a cereal bar with cranberries along with 250ml water, tested once, in different weeks, within 10-15min. Fingertip capillary blood glucose samples were taken at baseline, 15, 30, 45,60, 90 and 120min.
Other: Cocoa drink — Twelve healthy, normal weight subjects (male: 6,female: 6) after 10-14 hr fast, consumed 25g available carbohydrates from cocoa powder mixed with 500ml fat-free milk, tested once, in different weeks, within 5-10min. Fingertip capillary blood glucose samples were taken at baseline, 15, 30, 45,60, 90 and 120min.

SUMMARY:
This study investigated the effects of three commonly used sugar-free snacks with added sweeteners on glycemic responses

DETAILED DESCRIPTION:
This study aimed at 1. to determine the glycemic index and glycemic load of three sugar-free products with added sweeteners: apricot jam, cranberry cereal bar, and cocoa drink, and 2. to investigate the effects of these products on the postprandial glycemic response in healthy subjects

ELIGIBILITY:
Inclusion Criteria:

* healthy
* non-smoking
* non-diabetic men and women
* body mass index (BMI) between 18 and 29.9 kg/m2

Exclusion Criteria:

* severe chronic disease (e.g. coronary heart disease, diabetes mellitus,kidney or liver conditions, endocrine conditions)
* gastrointestinal disorders
* pregnancy
* lactation
* competitive sports
* alcohol
* drug dependency

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2020-07-30 (Actual); Primary Completion 2020-09-30 (Actual); Study Completion 2020-09-30 (Actual)

PRIMARY OUTCOMES:
Capillary blood glucose responses | 2 hours
  Clinically useful change in blood glucose, defined as the restoration of glucose within normal limits during the 2hr glucose tolerance test

SECONDARY OUTCOMES:
Subjective appetite ratings | 2 hours
  Useful change in subjective appetite using visual analogue scales with a score 0 to 10 (given in the form of booklet,one scale per page) at baseline, 15, 30, 45, 60, 90 and 120 min. The minimum or maximum score will be evaluated if it is better or worse depending on the appetite variable e.g hunger, satiety, desire to eat etc.

CONTACTS AND LOCATIONS:
Overall Officials: Aimilia Papakonstantinou, PhD, Principal Investigator — Agricultural University of Athens
Locations (1):
- Agricultural University of Athens, Athens, Attica, Greece